CLINICAL TRIAL: NCT07357922
Title: Association Between Maternal Serum Progesterone Levels and Threatened Abortion in Lactating Pregnant Women
Brief Title: Serum Progesterone and Threatened Abortion During Lactation
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Burak Deniz Aydoğdu, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 2025/517
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Threatened Abortion
Keywords: Serum Progesterone Levels; Threatened Abortion; Lactation During Pregnancy
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactating Pregnant Women (First Trimester): Pregnant women who conceived during the lactation period and are in the first trimester of pregnancy. Maternal serum progesterone levels will be measured at enrollment. Participants will be prospectively followed to evaluate the occurrence of threatened abortion, defined as first-trimester vaginal bleeding with a viable intrauterine pregnancy. This is a prospective observational cohort study, and no interventions are assigned.

SUMMARY:
This study aims to evaluate the effect of first-trimester maternal serum progesterone levels on threatened abortion in women who conceive during the lactation period. Serum progesterone concentrations will be measured in lactating pregnant women during the first trimester, and their association with the etiology of threatened abortion will be analyzed.

Threatened abortion is defined as vaginal bleeding occurring in the first trimester of pregnancy and represents a risk for early pregnancy loss. Previous studies have shown that serum progesterone levels may be lower in cases of threatened abortion compared to healthy pregnancies and play an essential role in predicting miscarriage risk. Serum progesterone is therefore considered a useful biomarker for assessing pregnancy viability and prognosis.

During lactation, progesterone levels may vary depending on breastfeeding duration and maternal hormonal status, and generally remain low, similar to follicular-phase levels in non-pregnant women. However, normal reference values during lactation are not well established. This study aims to contribute new data to the limited literature on the relationship between lactation, serum progesterone levels, and threatened abortion, and to provide insights that may help improve early pregnancy loss prevention strategies.

DETAILED DESCRIPTION:
This study is designed to investigate the relationship between maternal serum progesterone levels and threatened abortion in women who conceive during the lactation period. The primary objective is to evaluate first-trimester serum progesterone concentrations in lactating pregnant women and to assess their role in the etiology and clinical course of threatened abortion.

Threatened abortion is characterized by vaginal bleeding during the first trimester of pregnancy and is associated with an increased risk of early pregnancy loss. Progesterone plays a critical role in the maintenance of early pregnancy by supporting endometrial receptivity, suppressing uterine contractility, and modulating maternal immune tolerance. Previous studies have demonstrated that serum progesterone levels tend to be lower in pregnancies complicated by threatened abortion compared to uncomplicated pregnancies, and that reduced progesterone concentrations may be predictive of subsequent miscarriage.

Lactation is associated with distinct hormonal changes, primarily mediated by elevated prolactin levels, which suppress ovulation and result in progesterone levels comparable to those observed during the follicular phase of the menstrual cycle. Although progesterone levels increase following conception, the hormonal milieu during lactation may influence progesterone production and regulation in early pregnancy. However, normal reference ranges for serum progesterone levels in lactating pregnant women have not been clearly established, and data regarding their association with threatened abortion remain limited.

In this study, pregnant women who conceive during the lactation period will be enrolled. Maternal serum progesterone levels will be measured during the first trimester, and participants will be evaluated for the presence or absence of threatened abortion, defined as first-trimester vaginal bleeding with a viable intrauterine pregnancy. Clinical, obstetric, and demographic data will be recorded to allow assessment of potential confounding factors.

By examining the relationship between serum progesterone levels and threatened abortion in lactating pregnancies, this study aims to provide new insights into the hormonal mechanisms underlying early pregnancy complications. The findings may contribute to improved risk stratification, early diagnosis, and management strategies for threatened abortion in this specific population. Additionally, the study seeks to expand the limited body of literature on lactation-associated hormonal changes during early pregnancy and their clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 50 years.
* Pregnant women who conceived during the lactation period.
* Singleton pregnancy.
* First-trimester pregnancy.
* Availability of first-trimester serum progesterone measurement obtained as part of routine antenatal care.
* Ongoing follow-up at the participating hospitals.

Exclusion Criteria:

* Age under 18 years or over 50 years.
* Multiple pregnancies.
* Known chronic medical diseases.
* Use of progesterone supplementation before serum progesterone measurement.
* Missing or incomplete clinical or laboratory data.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is limited to individuals of female biological sex who are pregnant and in the lactation period.
Study Population: The study population consists of lactating pregnant women aged 18 to 50 years who present for routine antenatal care during the first trimester of pregnancy at the participating obstetrics and gynecology clinics. Eligible participants include women who conceived while breastfeeding and have available first-trimester serum progesterone measurements. Participants will be prospectively followed to evaluate the occurrence of threatened abortion and early pregnancy outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Threatened Abortion in Lactating Pregnant Women | From enrollment in the first trimester until 14 weeks of gestation
  The incidence of threatened abortion, defined as first-trimester vaginal bleeding with a viable intrauterine pregnancy, assessed by clinical evaluation and ultrasonographic confirmation.

SECONDARY OUTCOMES:
First-Trimester Serum Progesterone Levels | At enrollment during the first trimester of pregnancy
  Maternal serum progesterone levels measured during the first trimester of pregnancy will be recorded and compared between women with and without threatened abortion.
Early Pregnancy Loss | Up to 14 weeks of gestation
  The occurrence of pregnancy loss before 14 weeks of gestation will be recorded and evaluated in relation to first-trimester serum progesterone levels.
Serum Progesterone Cut-off Value for Predicting Threatened Abortion | During the first trimester of pregnancy
  The optimal first-trimester serum progesterone cut-off value for predicting threatened abortion in lactating pregnant women will be determined using receiver operating characteristic (ROC) curve analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Burak D. Aydoğdu, M.D., Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization

IPD SHARING:
Plan to Share IPD: No
Although data would be de-identified before any potential sharing, individual participant data will not be shared because the original ethics committee approval and informed consent do not permit data sharing beyond the study team. In addition, the dataset contains detailed clinical and laboratory variables that could carry a risk of re-identification. Any future data sharing would require additional ethics committee approval and updated participant consent. Study results will be disseminated in aggregated and anonymized form through scientific publications.

REFERENCES:
- [Background] Sammut L, Bezzina P, Gibbs V, Muscat-Baron Y, Agius-Camenzuli A, Calleja-Agius J. Predicting first-trimester pregnancy outcome in threatened miscarriage: A comparison of a multivariate logistic regression and machine learning models. Radiography (Lond). 2025 Oct;31(6):103159. doi: 10.1016/j.radi.2025.103159. Epub 2025 Sep 4. PMID 40912049
- [Background] Jiang TT, Zhang DY, Liu ZY, Lu ZS, Yan LM, Sun S, Xie JA, Zhu M, Zhang ZH, Wan YH, Wang H, Hao JH, Zhang C. Association of co-exposure to EDCs in early pregnancy with threatened abortion: The mediation effect of progesterone. Environ Int. 2025 Dec 11;207:110001. doi: 10.1016/j.envint.2025.110001. Online ahead of print. PMID 41391232